CLINICAL TRIAL: NCT04136730
Title: Effects of Home-based Resistance Exercise on Body Composition, Muscle Strength and Glycemic Control in People With Type 2 Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dasman Diabetes Institute (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr. Ebaa Al Ozairi, Chief Medical Officer, Dasman Diabetes Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM-2019-021
Record Dates: First submitted 2019-10-21; First posted 2019-10-23 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Home Care Services, Hospital-Based

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual Care
- Home-based (Active Comparator): Home-based resistance exercise training
  Interventions: Behavioral: Home-based

INTERVENTIONS:
Behavioral: Home-based — Resistance exercise carried out unsupervised at home
  Arms: Home-based

SUMMARY:
This study investigates the effects of home-based resistance exercise training, compared to a control group, on body composition, muscle strength and glycaemic control in people with type 2 diabetes.

Half participants will be in the home-based exercise group and half in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed type 2 diabetes
* No changes in anti-diabetic medication in the last 3 months

Exclusion Criteria:

* Not currently or in the past year participating in any vigorous aerobic activity (>1h per week) or any resistance exercise.
* BMI of 45 or higher
* Blood pressure of 160/100mmHg or higher
* Currently receiving insulin therapy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Glycated Haemoglobin concentration (mmol/mol) | Change from baseline to 32 weeks
  Glycated haemaglobin

SECONDARY OUTCOMES:
Fat-free mass | Change from baseline to 32 weeks
  Whole body fat free mass
Short performance physical battery test | Change from baseline to 32 weeks
  Short performance physical battery test (0 (worst performance) to 12 (best performance))

OTHER OUTCOMES:
Grip strength | Change from baseline to 32 weeks
  Grip strength measured by handheld dynamometer
One rep max | Change from baseline to 32 weeks
  The maximum weight that can be lifted for a single repetition of leg extension and lateral pull down
Push up test | Change from baseline to 32 weeks
  Number of push ups that can be performed
BMI | Change from baseline to 32 weeks
  Body mass index
Body fat | Change from baseline to 32 weeks
  Total body fat measured via DEXA
Visceral fat | Change from baseline to 32 weeks
  Visceral adipose tissue measured by DEXA
Physical activity levels | Change from baseline to 32 weeks
  Physical activity levels measured with a wrist worn accelerometer
Quality of life score | Change from baseline to 32 weeks
  EQ-5D-DL questionnaire will be used (5 (worst) to 125 (best))

CONTACTS AND LOCATIONS:
Overall Officials: Ebaa AlOzairi, Principal Investigator — Dasman Diabetes Institute
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al Ozairi E, Alsaeed D, Taliping D, Jalali M, El Samad A, Mashankar A, Taghadom E, Guess N, Gill JMR, Sattar N, Gray C, Welsh P, Gray SR. Protocol for a randomised controlled trial to investigate the effect of home- and gym-based resistance exercise training on glycaemic control, body composition and muscle strength. Trials. 2020 Jun 22;21(1):557. doi: 10.1186/s13063-020-04480-2. PMID 32571396